CLINICAL TRIAL: NCT03387579
Title: Comparison of Composite Lipid Emulsion Containing Fish Oil to Soy-based Lipid Reduction for Cholestasis Prevention in Neonates Requiring Abdominal Surgery
Brief Title: Comparison of Smoflipid to Soy-based Lipid Reduction for Cholestasis Prevention in Surgical Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Charles P.B. Vanderpool, Assistant Professor of Clinical Pediatrics, Co-chair, Nutrition Support Team at Riley Hospital for Children, Medical Director, Pediatric Intestinal Rehabilitation Program, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1708745276
Record Dates: First submitted 2017-12-03; First posted 2018-01-02 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Cholestasis of Parenteral Nutrition
MeSH Terms: interventions — SMOFlipid; Injections; soybean oil, phospholipid emulsion

STUDY DESIGN:
Intervention Model Description: Prospective patients will be randomized to one of the two treatment arms, either composite lipid containing fish oil (Smoflipid) or soy-based lipid reduction. A third arm will include retrospective patients who will act as controls and received soy-based lipid at standard dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Smoflipid 20% (Experimental): Patients randomized to this arm will receive the composite fish oil lipid, Smoflipid, at standard dosing up to 3 g/kg/day. Patients will be started on a dose of 1 g/kg/day and titrated up to maximum dose. As enteral nutrition is advanced the lipid dose will be weaned per study protocol and dietary recommendations.
  Interventions: Drug: Smoflipid 20% Lipid Emulsion for Injection
- Intralipid 20% Reduction (Experimental): Patients randomized to this arm will receive soy-based lipid (Intralipid) at a dose of 1 g/kg/day throughout their enrollment in the study.
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Intralipid 20% Historic (Other): Patients who retrospectively received soy-based lipid (Intralipid) at standard dosing of 2-3 g/kg/day were eligible for inclusion. Patients in this group were matched to prospective patients based on diagnosis, gestational age, and length of lipid therapy.
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion

INTERVENTIONS:
Drug: Smoflipid 20% Lipid Emulsion for Injection — Intravenous lipid containing soy, MCT, olive, and fish oils at goal doses of 3 g/kg/day
  Arms: Smoflipid 20%
Drug: Intralipid, 20% Intravenous Emulsion — Intravenous lipid emulsion of 20% soy oil at goal doses of 1 g/kg/day
  Other Names: Intralipid 20% Reduction
  Arms: Intralipid 20% Reduction
Drug: Intralipid, 20% Intravenous Emulsion — Intravenous lipid emulsion of 20% soy oil at goal doses of 2-3 g/kg/day
  Other Names: Intralipid 20% Historic
  Arms: Intralipid 20% Historic

SUMMARY:
Intestinal failure associated liver disease is a cholestatic liver disease associated with prolonged need for parenteral nutrition that can lead to such significant complications as liver failure. In the neonatal population, infants with history of intestinal resection and short bowel syndrome are at increased risk for this disease. The investigators plan to compare two possible lipid dosing preventative strategies including a composite, fish oil lipid and soy-based lipid reduction.

DETAILED DESCRIPTION:
Intestinal failure associated liver disease (IFALD) is a cholestatic liver disease associated with prolonged need for parenteral nutrition. This disease can lead to such serious complications as liver failure and need for transplantation. In the neonatal population, short bowel syndrome, due to intestinal resection, is the most common cause of intestinal failure. While the exact cause is yet to be determined, it is felt the lipid component of parenteral nutrition is a large contributor to the development of this disease. Currently, there is no standard preventative strategy to attempt to decrease the risk of IFALD in the high risk, post-surgical neonatal population. The investigators aim to complete a randomized trial comparing two possible preventative strategies. One group will receive a composite lipid containing fish oil (Smoflipid) and the other group will receive soy-based lipid at reduced dosing.

ELIGIBILITY:
Inclusion Criteria: Neonates with anticipated need for parenteral nutrition (based on primary physicians opinion) for greater than or equal to four weeks and one of the following diagnoses:

* Anatomic: Neonate with intestinal atresia, omphalocele, gastroschisis, or volvulus with or without intestinal resection.
* Ischemic/perforation: Neonates with spontaneous intestinal perforation or necrotizing enterocolitis requiring surgical intervention.

Exclusion Criteria:

* Current weight less than 750 grams
* AST or ALT greater than 5 times the upper limit of normal within 2 weeks of enrollment
* Direct bilirubin greater than 2 mg/dL on any consecutive measurements 5 - 7 days apart within 2 weeks of enrollment
* Severe coagulopathy with INR greater than 95th percentile for age (>1.7 at less than 5 days of age, > 1.5 older than five days of age)
* Culture confirmed sepsis with positive blood, urine, or CSF culture within 2 weeks of enrollment
* Renal failure requiring dialysis
* Cyanotic heart disease requiring prostaglandin therapy
* Hypertriglyceridemia (greater than 250mg/dL) at time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2024-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were eligible for enrollment if they were admitted to the level IV NICU, required abdominal surgery, and needed TPN. Patients were excluded if they had signs of liver disease at baseline. Informed consent was obtained, and once screening lab work completed patients were randomized into one of two prospective treatment groups. Historic controls were included from previous two years prior to enrollment with selection based on same eligibility criteria.
Pre-assignment Details: Screening labs including AST, ALT, GGT, platelet count, INR, and triglyceride level were performed prior to or at enrollment. Results were required prior to randomization. Only one patient was enrolled but found to have abnormal INR so was not randomized.
Groups:
- Smoflipid 20%: Smoflipid 20% is an intravenous lipid emulsions containing soy, MCT, olive, and fish oils. Patients randomized to this arm received the composite fish oil lipid, Smoflipid 20%, at dosing goal of 3 g/kg/day. Patients were started on a dose of 1 g/kg/day and titrated by 1g/kg/day up to goal. As enteral nutrition was advanced the lipid dose was weaned per study protocol and dietary recommendations.
  Smoflipid was infused over a 24 hour period, with infusion changed every 12 hours per hospital policy.
- Intralipid 20% Reduction: Intralipid 20% is an intravenous lipid emulsion containing soybean oil. Patients randomized to this arm received soy-based lipid (Intralipid 20%) at a goal dose of 1 g/kg/day. Lipid was increased incrementally by 0.5 g/kg/day every 3-5 days for growth less than goal of 25-30 g/kg/day despite maximization or remaining TPN components. Once adequate weight gain was established Intralipid was weaned back to goal of 1 g/kg/day by 0.5-1 g/kg/day increments. With enteral feeding advancement Intralipid was continued at 1 g/kg/day until TPN is stopped.
  Intralipid was infused over a 24 hour period, with infusion changed every 12 hours per hospital policy.
- Intralipid 20% Historic: A control group of historic patients who received Intralipid 20% at dosing of greater than or equal to 2 g/kg/day were included. Patients were enrolled using the same eligibility criteria as prospective patients.
  Given patients were retrospective, only available data in the patient electronic medical record was recorded.
Period: Overall Study
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Started | 12 | 12 | 24
Completed | 12 | 12 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic | Total
Number analyzed (Participants) | 12 | 12 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 4 [3.3 to 11.3] | 5 [4 to 5] | 2 [1 to 2.8] | 3.5 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 9 | 21
  Male | 5 | 7 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 11 | 12 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 8 | 10
  White | 10 | 11 | 13 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cholestasis
Description: Cholestasis was defined as a direct bilirubin > 2 mg/dL on two measurements 5 to 7 days apart.
Time Frame: Patients were monitored during time enrolled in study for a maximum of up to 12 weeks or 84 days.
Population: All participants who received study lipid or were included as historic controls.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
Participants | 1 | 3 | 7
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.590, Fisher Exact
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.224, Fisher Exact
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Weight Velocity
Description: Weight velocity was calculated as the difference in weight from end to start of study divided by number of days enrolled in study.
Time Frame: Patient weight was recorded at enrollment, weekly during time enrolled, and at end of study for up to a maximum of 12 weeks. End and enrollment weights were used to calculate velocity.
Population: All participants included.
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
grams per day | 28.6 (10.6) | 23.0 (11.9) | 24.6 (8.2)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.471, Kruskal-Wallis

3. Secondary Outcome: Length Velocity
Description: Length velocity was defined as the difference in length from end of study compared to enrollment divided by the number of days enrolled in study.
Time Frame: Length was measured at enrollment, weekly during time enrolled in study, and end of study up to a maximum of 12 weeks. End and enrollment measurements were used for velocity.
Measure: Mean (Standard Deviation); unit: centimeters per day
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
centimeters per day | 0.13 (0.08) | 0.09 (0.65) | 0.10 (0.08)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.525, Kruskal-Wallis

4. Secondary Outcome: Head Circumference (OFC) Velocity
Description: OFC velocity was calculated as difference end and start of study divided by number of days enrolled in study.
Time Frame: OFC was measured at enrollment, weekly, and end of study. Enrollment and end of study measurements used for velocity.
Measure: Mean (Standard Deviation); unit: centimeters per day
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
centimeters per day | 0.09 (0.03) | 0.07 (0.06) | 0.10 (0.05)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.753, Kruskal-Wallis

5. Secondary Outcome: Average Total Calorie Intake
Description: Total calorie intake, including parenteral and enteral sources, were averaged on a weekly basis.
Time Frame: Daily calorie intake was recorded and averaged on a weekly basis for duration of study enrollment up to max of 12 weeks.
Measure: Mean (Standard Deviation); unit: kcal per kilograms per day
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
kcal per kilograms per day | 114.0 (9.1) | 101.9 (10.5) | 109.1 (8.3)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.008, Kruskal-Wallis

6. Secondary Outcome: Number of Patients With Enteral Autonomy at End of Study
Description: Percentage of patients with enteral autonomy at time of leaving or stopping study was calculated. Enteral autonomy was defined as relying on enteral nutrition only for nutrition intake with no need for parenteral nutrition supplementation.
Time Frame: Enteral autonomy was recorded at the study end point for each individual patient. This end point was at time of stopping study lipid, discharge from hospital, or maximum of 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
Participants | 9 | 10 | 23
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.127, Fisher Exact

7. Secondary Outcome: Number of Patients With Essential Fatty Acid Deficiency (EFAD)
Description: Essential fatty acid deficiency was defined as a triene to tetraene ratio greater than 0.05.
Time Frame: Essential fatty acid levels were measured every 4 weeks during enrollment for a maximum of up to 12 weeks.
Population: Only prospective participants were included in this analysis as retrospective controls did not have essential fatty acid levels obtained.
Measure: Count of Participants; unit: Participants
Groups:
- Smoflipid 20%: Patients randomized to this arm will receive the composite fish oil lipid, Smoflipid, at standard dosing up to 3 g/kg/day. Patients will be started on a dose of 1 g/kg/day and titrated up to maximum dose. As enteral nutrition is advanced the lipid dose will be weaned per study protocol and dietary recommendations.
  Lipid Emulsions, Intravenous: Intravenous lipid containing soy, MCT, olive, and fish oils
- Intralipid 20% Reduction: Patients randomized to this arm will receive soy-based lipid (Intralipid) at a dose of 1 g/kg/day throughout their enrollment in the study.
  Intralipid, 20% Intravenous Emulsion: Intravenous lipid emulsion of 20% soy oil
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 12 | 12
Participants | 0 | 1
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 1.00, Fisher Exact

8. Secondary Outcome: AST Change Over Time
Description: The change of AST over time was calculated and compared between groups. AST change was calculated as AST end - AST enrollment.
Time Frame: AST was recorded at enrollment and every 2 weeks while enrolled in the study up to a maximum of 12 weeks.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
units per liter | -8.3 (25.5) | 2.9 (62.4) | 5.1 (49.8)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.046, Mixed Models Analysis — Intralipid 20% reduction versus smoflipid 20%; estimate = 8.553 — standard error 4.249
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.040, Mixed Models Analysis — Intralipid 20% historic versus smoflipid; estimate = 7.023 — standard error 3.376
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.718, Mixed Models Analysis — Intralipid 20% Historic versus Intralipid 20% reduction; estimate = -1.530 — standard error 4.231

9. Secondary Outcome: ALT Change Over Time
Description: The rate of change of ALT over time was compared between groups using mixed model analysis. Change of ALT was calculated as ALT at end of study compared to ALT at enrollment.
Time Frame: ALT measured at enrollment and every 2 weeks for max 12 weeks.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
units per liter | 8.7 (14.9) | 25.3 (53.3) | 17.2 (51.7)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.003, Mixed Models Analysis — Intralipid 20% reduction versus Smoflipid 20%; estimate = 13.436 — standard error 4.440
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.270, Mixed Models Analysis — Intralipid 20% historic versus Smoflipid 20%; estimate = 3.936 — standard error 3.553
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.034, Mixed Models Analysis — Intralipid 20% historic versus Intralipid 20% reduction; estimate = -9.500 — standard error 4.416

10. Secondary Outcome: Alkaline Phosphatase Change Over Time
Description: Alkaline phosphatase was recorded at enrollment and every 2 weeks. The change in alkaline phosphatase was calculated as alkaline phosphatase at end minus enrollment.
Time Frame: Alkaline phosphatase was measured at enrollment and every 2 weeks for max of 12 weeks.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
units per liter | 107.0 (146.9) | 166.1 (126.6) | 150.2 (139.9)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.006, Mixed Models Analysis — Intralipid 20% reduction versus Smoflipid 20%; estimate = 42.674 — standard error 15.216
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.305, Mixed Models Analysis — Intralipid 20% historic versus smoflipid 20%; estimate = 11.117 — standard error 10.771
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p < 0.001, Mixed Models Analysis — Intralipid 20% historic versus Intralipid 20% reduction; estimate = -31.557 — standard error 67.673

11. Secondary Outcome: Triglyceride Level Over Time
Description: All enrolled patients had serum triglyceride levels monitored at enrollment and weekly. The triglyceride level changes was calculated using values at the end of study compared to enrollment with mean and standard deviation calculated for each treatment group.
Time Frame: Serum triglyceride levels monitored at enrollment and weekly during time enrolled in study for a maximum of 12 weeks.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
mg/dL | -18.5 (31.0) | 013.3 (54.5) | 13.7 (48.0)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.835, Mixed Models Analysis — Intralipid 20% reduction versus smoflipid 20%; estimate = -0.593 — standard error 2.848
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.799, Mixed Models Analysis — Intralipid 20% historic versus smoflipid 20%; estimate = -0.522 — standard error 2.050
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.714, Mixed Models Analysis — Intralipid 20% historic versus Intralipid 20% reduction; estimate = 0.714 — standard error 2.758

12. Secondary Outcome: Gamma Glutamyl Transferase (GGT) Over Time
Description: GGT was documented at baseline and regularly intervals with level compared over time between groups. GGT was compared by treatment group for levels at end of study and enrollment.
Time Frame: GGT was measured at enrollment and every 2 weeks while enrolled in the study for a maximum of up to 12 weeks.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
units per liter | -0.8 (99.7) | 55.7 (73.3) | 37.3 (121.7)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.379, Mixed Models Analysis; Intralipid 20% reduction versus smoflipid 20%; estimate = 11.162 — standard error 12.626
Statistical Analysis 2: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 0.717, Mixed Models Analysis — Intralipid 20% historic versus smoflipid 20%; estimate = 3.853 — standard error 10.615
Statistical Analysis 3: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority — Intralipid 20% historic versus intralipid 20% reduction; p = 0.576, Mixed Models Analysis; estimate = -7.310 — standard error 13.025

13. Secondary Outcome: Number of Patients With Retinopathy of Prematurity
Description: The rate of retinopathy of prematurity (ROP) was compared between groups. ROP was diagnosed based on ophthalmologist examination with all stages included.
Time Frame: Diagnosis was based on diagnosis during time of initial hospitalization to level 4 NICU.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
Participants | 2 | 1 | 3
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; ROP; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; ROP; Test type: Superiority; p = 1.00, Fisher Exact

14. Secondary Outcome: Number of Patients With Bronchopulmonary Dysplasia (BPD) or Chronic Lung Disease
Description: The rate of BPD was documented and compared between groups. BPD was diagnosed based on need for respiratory support at 28 days of age. All levels of severity were included.
Time Frame: All patient had diagnosis of BPD documented from admission at level 4 NICU.
Measure: Count of Participants; unit: Participants
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
Participants | 2 | 2 | 5
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.640, Fisher Exact
Statistical Analysis 3: Comparison: Smoflipid 20% vs Intralipid 20% Historic; Test type: Superiority; p = 1.00, Fisher Exact

15. Secondary Outcome: NICU Length of Stay
Description: The length of stay at the level 4 NICU was compared between groups.
Time Frame: Length of stay will be calculated based on documenting each patient's admission date and date leaving the NICU.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction | Intralipid 20% Historic
Number analyzed (Participants) | 12 | 12 | 24
days | 72.2 (57.6) | 33.3 (46.0) | 40.2 (42.2)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction vs Intralipid 20% Historic; Test type: Superiority; p = 0.211, Kruskal-Wallis

16. Secondary Outcome: Three Year Development- Communication
Description: During the third year of chronological age an Ages and Stages questionnaire (ASQ) was completed by the parents. For each section the range of score possible is 0-60. Higher scores show improved outcomes. Scores are separated into on schedule, monitoring zone, and below cutoff. These thresholds vary by aged screened. Possible screens used for this age group include 36 months, 42 months, and 48 months dependent on exact chronologic age screen completed. At 36 months communication 45-60 is on schedule; 35-40 monitoring, and <35 below cutoff. For 42 months on schedule 40-60; monitoring 30-35; below cutoff <35. For 48 months on schedule 45-60; monitoring 35-40; below cutoff <35.
Time Frame: ASQ was completed during the third year of life from 3 years 0 days to 3 years 364 days of chronologic age.
Population: Only the prospective patients treated by the research team were included in developmental assessment. The Intralipid 20% Historic group was not included in analysis as these patients were not treated by the research team and developmental screening could not be performed on these patients. Data for the "Intralipid 20% Historic" arm was not collected as specified by the study protocol and statistical analysis plan.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 10 | 10
score on a scale | 40.3 (22.4) | 41.2 (17.7)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.720, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Three Year Development: Gross Motor
Description: During the third year of chronological age an Ages and Stages questionnaire (ASQ) was completed by the parents. For each section the range of score possible is 0-60. Higher scores indicate improved outcome, there are three possible scoring categories on schedule (normal), monitoring zone, below cutoff. Score thresholds by possible screens include: 36 months on schedule 50-60; monitoring 40-45; below cutoff <40. 42 months on schedule 50-60; monitoring 40-45; below cutoff <40. 48 months on schedule 45-60; monitoring 35-40; below cutoff <35.
Time Frame: three year chronological age 3 years and 0 days to 3 years and 364 days
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 10 | 10
score on a scale | 43.0 (24.2) | 54.1 (8.19)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.500, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Three Year Development: Fine Motor
Description: During the third year of chronological age an Ages and Stages questionnaire (ASQ) was completed by the parents. For each section the range of score possible is 0-60. Higher scores show improved outcomes with three scoring categories: on schedule (normal), monitoring zone, and below cutoff. These thresholds vary by each category and screening age. Based on the possible screens for chronological age the score categories are: 36 months: 35-60 on schedule; 20-30 monitoring; <20 below cutoff. 42 months: 35-60 on schedule; 20-30 monitoring; <20 below cutoff. 48 months: 35-60 on schedule; 20-30 monitoring; <20 below cutoff.
Time Frame: three year chronological age (3 years and 0 days to 3 years and 364 days)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 10 | 10
score on a scale | 32.2 (21.6) | 34.9 (19.1)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.774, t-test, 2 sided

19. Secondary Outcome: Three Year Development: Problem Solving
Description: During the third year of chronological age an Ages and Stages questionnaire (ASQ) was completed by the parents. For each section the range of score possible is 0-60. Higher scores indicate improved outcomes with three possible score categories: on schedule (normal), monitoring zone, and below cutoff. Category thresholds vary by outcome category and age of screen. There are three possible screens that were used for this population, chosen based on chronologic age. The score categories based on age are: 36 months: 45-60 on schedule; 35-40 monitoring; <35 below cutoff. 42 months: 40-60 on schdule; 30-35 monitoring; <30 below cutoff. 48 months: 45-60 on schedule; 35-40 monitoring; <35 below cutoff
Time Frame: three year chronological age (3 years and 0 days to 3 years and 364 days)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 10 | 10
score on a scale | 47.9 (19.5) | 47.3 (11.1)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.457, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Three Year Development: Personal Social
Description: During the third year of chronological age an Ages and Stages questionnaire (ASQ) was completed by the parents. For each section the range of score possible is 0-60. Higher scores indicate improved outcomes with three score categories possible including on schedule (normal), monitoring zone, and below cutoff. These thresholds vary based on outcome measure and age of screen completed. Screen used depends on chronological age at screen. Score thresholds for each age include: 36 months: 45-60 on schedule; 35-40 monitoring; <35 below cutoff. 42 months: 45-60 on schedule; 35-40 monitoring; <35 below cutoff. 48 months: 40-60 on schedule; 30-40 monitoring; <30 below cutoff.
Time Frame: three year chronological age (3 years and 0 days to 3 years and 364 days)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
Number analyzed (Participants) | 10 | 10
score on a scale | 46.5 (20.6) | 47.1 (10.5)
Statistical Analysis 1: Comparison: Smoflipid 20% vs Intralipid 20% Reduction; Test type: Superiority; p = 0.475, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while patient was receiving study lipid, up to a maximum of 12 weeks.
Description: Adverse event data was not collected during the retrospective analysis of the historical control arm (Intralipid 20% Historic).
Groups:
- Smoflipid 20%: Patients randomized to this arm received the composite fish oil lipid, Smoflipid, at standard dosing up to 3 g/kg/day. Patients started on a dose of 1 g/kg/day and titrated up to maximum dose. As enteral nutrition was advanced the lipid dose was weaned per study protocol and dietary recommendations.
- Intralipid 20% Reduction: Patients randomized to this arm received soy-based lipid (Intralipid) at a dose of 1 g/kg/day throughout their enrollment in the study.
Arm/Group | Smoflipid 20% | Intralipid 20% Reduction
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12 | 2/12
Other Adverse Events (participants affected / at risk) | 8/12 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoflipid 20% (N=12) | Intralipid 20% Reduction (N=12)
Rapid infusion (Product Issues) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoflipid 20% (N=12) | Intralipid 20% Reduction (N=12)
Elevated GGT (Gastrointestinal disorders) | 1 (1) | 2 (2) — GGT documented at enrollment and weekly.
Elevated LFT (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 8 (15) | 6 (12) — Anemia was defined based on set hematocrit parameters.
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochloremia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperchloremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Essential fatty acid deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Elevated magnesium (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased respiratory support (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Elevated alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Feeding intolerance (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03387579/Prot_SAP_002.pdf